CLINICAL TRIAL: NCT05325723
Title: Evaluation of an Automated Smartphone-based Digital Auscultation Application for Detecting Abnormal Heart Sounds Using Deep Learning Techniques - the Automated Valvular Heart Disease Assessment (AVDA) Pilot Study
Brief Title: Evaluation of an Automated Smartphone-based Digital Auscultation Application for Detecting Abnormal Heart Sounds Using Deep Learning Techniques
Acronym: AVDA
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02515; am21Eckstein
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Valvular Heart Disease
Keywords: automated digital auscultation; deep learning technique; smartphone-based digital auscultation; Computer-assisted auscultation (CAA); artificial neural networks (ANN); heart sound (HS) identification; medical grade audio phonocardiogram (PCG)
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention group: 1. 30 second audio phonocardiogram (PCG) recordings at each of the five standard cardiac auscultatory positions using an Apple iPhone®.
  2. the assessment of VHD by echocardiogram, as reported by the echocardiography laboratory.

SUMMARY:
This pilot study is to investigate the feasibility of obtaining medical grade audio phonocardiogram (PCG) recordings using a smartphone-based auscultation device in the first step. The ability to determine Valvular Heart Disease (VHD) (i.e., presence or absence of cardiac murmurs) using novel handheld CAA-devices shall be analyzed and first data on a smartphone-based auscultation in a hospital setting shall be collected. In further studies, the data provided from this study can be used to investigate the potential diagnostic use of such devices in the ambulatory and stationary care scenarios.

DETAILED DESCRIPTION:
Cardiac auscultation is considered to be highly subjective with substantial varying sensitivities and specificities in regard of the practitioners' expertise. Computer-assisted auscultation (CAA) aims to provide increased objectivity. CAA makes auscultation procedure less operator-dependent, approximate inter-examiner differences and may reduce uncertainties in the course of the examination. With the introduction of modern Machine Learning software libraries and ever-growing computational resources CAA has advanced significantly and is now able to classify heart sounds and murmurs into normal and abnormal, using complex spectro-temporal signal processing techniques and neural network pathways. CAA has simultaneously made the shift from the deployment on computers to consumer smartphones. A benefit of CAA can be expected from the smartphone alone in terms of cost, application range, the clinical validity of such algorithms should now be measured in this pilot study. This pilot study is to investigate the feasibility of obtaining medical grade audio phonocardiogram (PCG) recordings using a smartphone-based auscultation device in the first step. In further studies, the data provided from this study can be used to investigate the potential diagnostic use of such devices in the ambulatory and stationary care scenarios.

ELIGIBILITY:
Inclusion Criteria:

* Older or equal than 18 years of age
* Referred for an echocardiogram
* Able to provide informed consent

Exclusion Criteria:

* Confirmed arrythmia
* Prior valvular intervention
* Evidence of congenital heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at the Department of Cardiology, University Hospital Basel. The scheduled appointment lists of patients for an echocardiography will be checked and eligible patients will be contacted by the study physician before presenting for their planned echocardiography appointment.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Determination of Valvular Heart Disease (VHD) (i.e., presence or absence of cardiac murmurs) | one time assessment at baseline (approx. 5 minutes)
  Ability to determine VHD (i.e., presence or absence of cardiac murmurs) using novel handheld CAA-devices is investigated by collection of data on a smartphone-based auscultation in a hospital setting.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, Prof. Dr. med., Principal Investigator — University Hospital Basel, Division of Internal Medicine
Locations (1):
- University Hospital Basel, Division of Internal Medicine, Basel, Switzerland